CLINICAL TRIAL: NCT02559557
Title: Adaptation and Pilot-Testing a Parenting Intervention for Spanish-Speaking Parents of Children at Risk for Neurocognitive Late Effects
Brief Title: Culturally Adapted Parenting Intervention for Spanish-Speaking Parents in Improving Outcomes of Younger Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia Survivors at Risk for Late Neurocognitive Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15297; NCI-2015-01567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15297 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Cancer Survivor; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Cognitive Side Effects of Cancer Therapy
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (Spanish-adapted skills training) (Experimental): PHASE I (FOCUS GROUPS): Parents undergo a semi-structured interview with bilingual research assistants over 120 minutes. The content and purpose of the intervention is explained, and the focus group discussions elicit feedback on the intervention components and content of the sessions, and whether the material is culturally and linguistically appropriate. Following the focus group discussion, parents receive a copy of the educational handouts that they may choose to use with their child if they like.
  PHASE II (PILOT TESTING): Parents of children age 5 to 17 years, 11 months old undergo adapted skills training in Spanish over 60 minutes (8 training sessions total) or 80 minutes (6 training sessions total). The adapted skills training sessions focus on parenting strategies and learning techniques. Sessions include homework assignments and techniques for parents to apply with their child for at least 30 minutes, 3 times a week at home.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Participate in focus groups
  Other Names: Education for Intervention; Intervention, Educational
Other: Educational Intervention — Undergo Spanish-adapted skills training and homework assignments
  Other Names: Education for Intervention; Intervention, Educational
Other: Quality-of-Life Assessment — Answer questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Answer questionnaires

SUMMARY:
This pilot clinical trial studies a culturally adapted skills training and educational intervention in guiding parents of younger acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML) survivors at risk for long-term attention and memory problems (late neurocognitive effects). ALL and AML treatments target the central nervous system and may put younger survivors at increased risk for late neurocognitive effects, which may lead to learning difficulties or behavior problems and poor health-related quality of life. Spanish-speaking parents of young ALL or AML survivors may not have access to the information, resources, or guidance to help their children through these difficulties. Adapting an existing parent-training program into Spanish may help teach Spanish-speaking parents effective ways to prevent or reduce learning and behavioral difficulties, which may improve the quality of life of parents and young ALL or AML survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To culturally modify and adapt an existing educational and skills-training intervention for use with Spanish-speaking parents of children with acute lymphoblastic leukemia (ALL) or with acute myeloid leukemia (AML).

II. To pilot the culturally-modified, parenting intervention with eligible families of children treated for ALL or AML in the Pediatrics department at City of Hope.

OUTLINE:

PHASE I (FOCUS GROUPS): Parents undergo a semi-structured interview with bilingual research assistants over 120 minutes. The content and purpose of the intervention is explained, and the focus group discussions elicit feedback on the intervention components and content of the sessions, and whether the material is culturally and linguistically appropriate. Following the focus group discussion, parents receive a copy of the educational handouts that they may choose to use with their child if they like.

PHASE II (PILOT TESTING): Parents of children age 5 to 17 years, 11 months old undergo adapted skills training in Spanish over 60 minutes (8 training sessions total) or 80 minutes (6 training sessions total). The adapted skills training sessions focus on parenting strategies and learning techniques. Sessions include homework assignments and techniques for parents to apply with their child for at least 30 minutes, 3 times a week at home.

After completion of study, parents are followed up every 2 weeks for 3 months and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR FOCUS GROUPS (PHASE I)

* Parents or adult primary caregiver (e.g., grandmother) of children ages 5 to 17 in treatment remission and has completed intensive therapy for ALL or AML
* Parents of childhood cancer survivors who are now 18 years or older and who were previously treated for ALL or AML (do not need to live with the child)
* One or both of the parents will self-identify as Hispanic/Latino, the primary participating parent will be either Spanish speaking, bilingual, or is bilingual but identifies their primary language as English and will live with the child

INCLUSION CRITERIA FOR PILOT-TESTING (PHASE II)

* Parent/Caregiver: parents or adult primary caregiver (e.g., grandmother) of children treated for ALL or AML
* Parent/Caregiver: one or both of the parents will self-identify as Hispanic/Latino, the primary participating parent will be either Spanish speaking, bilingual, or is bilingual but identifies their primary language as English and will live with the child
* Child: child is in treatment remission and has completed intensive therapy
* Child: child is age 5 to 17 years, 11 months
* Child: child understands English

Exclusion Criteria:

EXCLUSION CRITERIA FOR FOCUS GROUPS (PHASE I)

* Parents of ALL or AML survivors with a history of a major psychiatric condition that precludes participation (e.g., psychosis, severe depression, active substance abuse)
* Existing history of severe cognitive impairment in the child as reported by the parents or documented in the child's City of Hope medical records

EXCLUSION CRITERIA FOR PILOT TESTING (PHASE II)

* Parent/Caregiver: parents with a history of a major psychiatric condition that precludes participation (e.g., psychosis, severe depression, active substance abuse)
* Child: survivors with a history of a major psychiatric condition that precludes participation (e.g., psychosis, severe depression, active substance abuse)
* Child: existing history of severe cognitive impairment (intelligence quotient [IQ] =< 70) as reported by the parents or the child's City of Hope medical records, or by the child's performance score on the Wechsler Intelligence Scale for Children (WISC) Working Memory and Processing Speed index measures administered in this study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-22; Primary Completion 2016-04-18 (Actual); Study Completion 2016-04-18 (Actual)

PRIMARY OUTCOMES:
Feasibility, measured by the percentage of parents who complete the entire adapted skills-training parenting intervention | After 6 sessions (up to 12 months)
  Feasibility will be operationally defined as > 75% of parents completing the intervention.

SECONDARY OUTCOMES:
Change in child's school-related health-related quality of life (HRQOL) score as assessed by the Pediatric Quality of Life scale | Baseline to up to 12 months
  Explored for pre- and post-intervention changes using descriptive analyses.
Change in learning strategies as measured by the School Motivation and Learning Strategies Inventory | Baseline to up to 12 months
  Explored for pre- and post-intervention changes using descriptive analyses.
Change in parent knowledge and efficacy, as measured by the Parent Knowledge, Beliefs, and Behaviors Questionnaire (PBQ) | Baseline to up to 12 months
  Explored for pre- and post-intervention changes using descriptive analyses.
Parent satisfaction with the intervention as measured by the perceived benefits scale | Up to 12 months
  Satisfaction with intervention is defined as group mean rating of > 3/5 on the perceived benefit scale. Perceived benefit will be examined using group means obtained from parents' ratings on satisfaction and barriers questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Patel, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States